CLINICAL TRIAL: NCT04166513
Title: Effects of tDCS in Language Recovery and Reorganization in Chronic Aphasia
Brief Title: Effects of Transcranial Direct Current Stimulation (tDCS) on Language
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Sara Pillay, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 33162
Record Dates: First submitted 2019-11-08; First posted 2019-11-18 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Aphasia
Keywords: tDCS; treatment; brain stimulation
MeSH Terms: conditions — Stroke; Aphasia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Partial crossover design. Participants will maintain one of two speech therapy modalities throughout the study, but will crossover from targeted to active control stimulation (or vice versa).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Care provider, participant, and outcome assessor are masked for tDCS status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (4):
- Targeted tDCS with Phonologic-Focused Speech Therapy (Experimental): Participants will receive phonologic-focused speech therapy with targeted anodal-tDCS for 10 therapy sessions before.
  Interventions: Device: Targeted Transcranial Direct Current Stimulation; Behavioral: Phonologic-Focused Speech Therapy
- Active Control tDCS with Phonologic-Focused Speech Therapy (Active Comparator): Participants will receive phonologic-focused speech therapy with active control tDCS for 10 therapy sessions.
  Interventions: Device: Active Control Transcranial Direct Current Stimulation; Behavioral: Phonologic-Focused Speech Therapy
- Targeted tDCS with Semantic-Focused Speech Therapy (Experimental): Participants will receive semantic-focused speech therapy with targeted anodal-tDCS for 10 therapy sessions.
  Interventions: Device: Targeted Transcranial Direct Current Stimulation; Behavioral: Semantic-Focused Speech Therapy
- Active Control tDCS with Semantic-Focused Speech Therapy (Active Comparator): Participants will receive semantic-focused speech therapy with active control tDCS for 10 therapy sessions.
  Interventions: Device: Active Control Transcranial Direct Current Stimulation; Behavioral: Semantic-Focused Speech Therapy

INTERVENTIONS:
Device: Targeted Transcranial Direct Current Stimulation — High-Definition-tDCS will be delivered via a battery-driven constant direct current stimulator (Soterix) using a 4x1 montage (1 central anodal electrode and 4 cathodal electrodes) arranged in a HD-cap. The current is turned on and increased in a ramplike fashion over approximately 30 seconds until reaching a strength of no more than 2mA, with a current density equal to 0.08mA/cm2. Stimulation will be maintained no longer than 20 minutes, and stimulation will be applied to the targeted region.
  Other Names: HD-tDCS; tDCS
  Arms: Targeted tDCS with Phonologic-Focused Speech Therapy; Targeted tDCS with Semantic-Focused Speech Therapy
Device: Active Control Transcranial Direct Current Stimulation — High-Definition-tDCS will be delivered via a battery-driven constant direct current stimulator (Soterix) using a 4x1 montage (1 central anodal electrode and 4 cathodal electrodes) arranged in a HD-cap. The current is turned on and increased in a ramplike fashion over approximately 30 seconds until reaching a strength of no more than 2mA, with a current density equal to 0.08mA/cm2. Stimulation will be maintained no longer than 20 minutes, and stimulation will be applied to the active control region.
  Other Names: Active Control tDCS; Active Control HD-tDCS
  Arms: Active Control tDCS with Phonologic-Focused Speech Therapy; Active Control tDCS with Semantic-Focused Speech Therapy
Behavioral: Phonologic-Focused Speech Therapy — Participants are asked to generate or choose from a list phonologic information about a target picture.
  Other Names: Phonologic Component Analysis
  Arms: Active Control tDCS with Phonologic-Focused Speech Therapy; Targeted tDCS with Phonologic-Focused Speech Therapy
Behavioral: Semantic-Focused Speech Therapy — Participants who have difficulty retrieving an object name are given hierarchical clues or asked questions about the objects function as a way of activating the semantic network for that object, leading to eventual retrieval of the target word.
  Other Names: Semantic Feature Analysis
  Arms: Active Control tDCS with Semantic-Focused Speech Therapy; Targeted tDCS with Semantic-Focused Speech Therapy

SUMMARY:
This study will investigate the effects of mild electrical stimulation in conjunction with speech therapy for people with post-stroke aphasia to enhance language recovery.

DETAILED DESCRIPTION:
Aphasia is a disturbance of language, primarily caused by brain injury to the left cerebral hemisphere. Aphasia treatments include speech and language therapy and pharmacologic therapy, but several studies have found that these treatments are not completely effective for patients with aphasia, leaving them with residual deficits that significantly add to the cost of stroke-related care. Additionally, the amount and frequency of speech and language therapy delivered may have a critical effect on recovery. Therefore, there is a need for new treatments or adjuncts to existing treatments, such as brain stimulation interventions, that have the potential to show greater improvements in patients with aphasia. One such new approach for non-invasive brain stimulation is transcranial direct current stimulation (tDCS).

This study will examine the effects of tDCS during speech therapy to further examine which method or methods is best for patient recovery. Patients enrolled in the study will undergo language testing that covers a broad range of language functions. Functional Magnetic Resonance Imaging (fMRI) will be completed before and after speech therapy intervention arms to investigate the neural processes affected by tDCS and speech therapy.

Study design:

Patients will be randomly assigned to one of 2 speech therapy groups in a double-blind, partial crossover design. Patients will receive one of two different speech therapy treatment interventions to focus on specific processing deficits. Participants will undergo neuropsychological evaluation and fMRI assessment before receiving targeted or active-control anodal-tDCS for 10 therapy sessions. Participants will then be re-tested using the behavioral assessment measure and fMRI before crossing over to either receive the tDCS intervention they did not already receive, within the same speech therapy arm. They will complete a behavioral assessment and fMRI at 3 months post Treatment 2 and a final behavioral assessment at 6 months post Treatment 2.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a language deficit from focal neurologic damage (e.g. stroke, tumor).
* Patients must be adults and have English-language fluency.
* Patients must be eligible to undergo MRI.

Exclusion Criteria:

* Advanced neurodegenerative disease (i.e. Stage 3 Alzheimer's disease) or neurologic disorder (e.g. idiopathic epilepsy, Parkinson's disease, ALS)
* Severe psychopathology (e.g. schizophrenia, bipolar disorder, acute major depressive episode)
* No suspected or diagnosed uncorrectable hearing or vision difficulties, or developmental disabilities (i.e. intellectual disability or learning disability).
* Contraindications to MRI such as claustrophobia, implanted electronic devices, MRI-incompatible metal in the body, extreme obesity, pregnancy, inability to lie flat, and inability to see or hear stimulus materials

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Pillay, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jordan LC, Hillis AE. Disorders of speech and language: aphasia, apraxia and dysarthria. Curr Opin Neurol. 2006 Dec;19(6):580-5. doi: 10.1097/WCO.0b013e3280109260. PMID 17102697
- [Background] Greener J, Enderby P, Whurr R. Pharmacological treatment for aphasia following stroke. Cochrane Database Syst Rev. 2001;2001(4):CD000424. doi: 10.1002/14651858.CD000424. PMID 11687079
- [Background] Brady MC, Kelly H, Godwin J, Enderby P. Speech and language therapy for aphasia following stroke. Cochrane Database Syst Rev. 2012 May 16;(5):CD000425. doi: 10.1002/14651858.CD000425.pub3. PMID 22592672
- [Background] Lincoln NB, McGuirk E, Mulley GP, Lendrem W, Jones AC, Mitchell JR. Effectiveness of speech therapy for aphasic stroke patients. A randomised controlled trial. Lancet. 1984 Jun 2;1(8388):1197-200. doi: 10.1016/s0140-6736(84)91690-8. PMID 6202993
- [Background] Ellis C, Simpson AN, Bonilha H, Mauldin PD, Simpson KN. The one-year attributable cost of poststroke aphasia. Stroke. 2012 May;43(5):1429-31. doi: 10.1161/STROKEAHA.111.647339. Epub 2012 Feb 16. PMID 22343643
- [Background] Ellis C, Dismuke C, Edwards KK. Longitudinal trends in aphasia in the United States. NeuroRehabilitation. 2010;27(4):327-33. doi: 10.3233/NRE-2010-0616. PMID 21160122
- [Background] Boysen AE, Wertz RT. Clinician Costs in Aphasia Treatment: How Much Is a Word Worth? Clin. Aphasiology 1996;24:207-213.
- [Background] Meinzer M, Djundja D, Barthel G, Elbert T, Rockstroh B. Long-term stability of improved language functions in chronic aphasia after constraint-induced aphasia therapy. Stroke. 2005 Jul;36(7):1462-6. doi: 10.1161/01.STR.0000169941.29831.2a. Epub 2005 Jun 9. PMID 15947279
- [Background] Holland R, Crinion J. Can tDCS enhance treatment of aphasia after stroke? Aphasiology. 2012 Sep;26(9):1169-1191. doi: 10.1080/02687038.2011.616925. Epub 2011 Nov 3. PMID 23060684
- [Background] Paulus W. Transcranial direct current stimulation (tDCS). Suppl Clin Neurophysiol. 2003;56:249-54. doi: 10.1016/s1567-424x(09)70229-6. PMID 14677402
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] Nitsche MA, Paulus W. Sustained excitability elevations induced by transcranial DC motor cortex stimulation in humans. Neurology. 2001 Nov 27;57(10):1899-901. doi: 10.1212/wnl.57.10.1899. PMID 11723286
- [Background] Liebetanz D, Nitsche MA, Tergau F, Paulus W. Pharmacological approach to the mechanisms of transcranial DC-stimulation-induced after-effects of human motor cortex excitability. Brain. 2002 Oct;125(Pt 10):2238-47. doi: 10.1093/brain/awf238. PMID 12244081
- [Background] Hamilton RH, Chrysikou EG, Coslett B. Mechanisms of aphasia recovery after stroke and the role of noninvasive brain stimulation. Brain Lang. 2011 Jul;118(1-2):40-50. doi: 10.1016/j.bandl.2011.02.005. Epub 2011 Apr 2. PMID 21459427
- [Background] Darkow R, Martin A, Wurtz A, Floel A, Meinzer M. Transcranial direct current stimulation effects on neural processing in post-stroke aphasia. Hum Brain Mapp. 2017 Mar;38(3):1518-1531. doi: 10.1002/hbm.23469. Epub 2016 Nov 11. PMID 27859982
- [Background] Meinzer M, Jahnigen S, Copland DA, Darkow R, Grittner U, Avirame K, Rodriguez AD, Lindenberg R, Floel A. Transcranial direct current stimulation over multiple days improves learning and maintenance of a novel vocabulary. Cortex. 2014 Jan;50:137-47. doi: 10.1016/j.cortex.2013.07.013. Epub 2013 Aug 6. PMID 23988131
- [Background] Reis J, Schambra HM, Cohen LG, Buch ER, Fritsch B, Zarahn E, Celnik PA, Krakauer JW. Noninvasive cortical stimulation enhances motor skill acquisition over multiple days through an effect on consolidation. Proc Natl Acad Sci U S A. 2009 Feb 3;106(5):1590-5. doi: 10.1073/pnas.0805413106. Epub 2009 Jan 21. PMID 19164589
- [Background] Cohen Kadosh R, Soskic S, Iuculano T, Kanai R, Walsh V. Modulating neuronal activity produces specific and long-lasting changes in numerical competence. Curr Biol. 2010 Nov 23;20(22):2016-20. doi: 10.1016/j.cub.2010.10.007. Epub 2010 Nov 4. PMID 21055945
- [Background] Vestito L, Rosellini S, Mantero M, Bandini F. Long-term effects of transcranial direct-current stimulation in chronic post-stroke aphasia: a pilot study. Front Hum Neurosci. 2014 Oct 14;8:785. doi: 10.3389/fnhum.2014.00785. eCollection 2014. PMID 25352798
- [Background] Gandiga PC, Hummel FC, Cohen LG. Transcranial DC stimulation (tDCS): a tool for double-blind sham-controlled clinical studies in brain stimulation. Clin Neurophysiol. 2006 Apr;117(4):845-50. doi: 10.1016/j.clinph.2005.12.003. Epub 2006 Jan 19. PMID 16427357
- [Background] Bikson M, Datta A, Elwassif M. Establishing safety limits for transcranial direct current stimulation. Clin Neurophysiol. 2009 Jun;120(6):1033-4. doi: 10.1016/j.clinph.2009.03.018. Epub 2009 Apr 24. No abstract available. PMID 19394269
- [Background] Iyer MB, Mattu U, Grafman J, Lomarev M, Sato S, Wassermann EM. Safety and cognitive effect of frontal DC brain polarization in healthy individuals. Neurology. 2005 Mar 8;64(5):872-5. doi: 10.1212/01.WNL.0000152986.07469.E9. PMID 15753425
- [Background] Brunoni AR, Amadera J, Berbel B, Volz MS, Rizzerio BG, Fregni F. A systematic review on reporting and assessment of adverse effects associated with transcranial direct current stimulation. Int J Neuropsychopharmacol. 2011 Sep;14(8):1133-45. doi: 10.1017/S1461145710001690. Epub 2011 Feb 15. PMID 21320389
- [Background] Monti A, Ferrucci R, Fumagalli M, Mameli F, Cogiamanian F, Ardolino G, Priori A. Transcranial direct current stimulation (tDCS) and language. J Neurol Neurosurg Psychiatry. 2013 Aug;84(8):832-42. doi: 10.1136/jnnp-2012-302825. Epub 2012 Nov 8. PMID 23138766
- [Background] Monti A, Cogiamanian F, Marceglia S, Ferrucci R, Mameli F, Mrakic-Sposta S, Vergari M, Zago S, Priori A. Improved naming after transcranial direct current stimulation in aphasia. J Neurol Neurosurg Psychiatry. 2008 Apr;79(4):451-3. doi: 10.1136/jnnp.2007.135277. Epub 2007 Dec 20. PMID 18096677
- [Background] Baker JM, Rorden C, Fridriksson J. Using transcranial direct-current stimulation to treat stroke patients with aphasia. Stroke. 2010 Jun;41(6):1229-36. doi: 10.1161/STROKEAHA.109.576785. Epub 2010 Apr 15. PMID 20395612
- [Background] Fiori V, Coccia M, Marinelli CV, Vecchi V, Bonifazi S, Ceravolo MG, Provinciali L, Tomaiuolo F, Marangolo P. Transcranial direct current stimulation improves word retrieval in healthy and nonfluent aphasic subjects. J Cogn Neurosci. 2011 Sep;23(9):2309-23. doi: 10.1162/jocn.2010.21579. Epub 2010 Oct 14. PMID 20946060
- [Background] Fridriksson J. Measuring and inducing brain plasticity in chronic aphasia. J Commun Disord. 2011 Sep-Oct;44(5):557-63. doi: 10.1016/j.jcomdis.2011.04.009. Epub 2011 Apr 30. PMID 21620414
- [Background] Marangolo P, Marinelli CV, Bonifazi S, Fiori V, Ceravolo MG, Provinciali L, Tomaiuolo F. Electrical stimulation over the left inferior frontal gyrus (IFG) determines long-term effects in the recovery of speech apraxia in three chronic aphasics. Behav Brain Res. 2011 Dec 1;225(2):498-504. doi: 10.1016/j.bbr.2011.08.008. Epub 2011 Aug 12. PMID 21856336
- [Background] Meinzer M, Darkow R, Lindenberg R, Floel A. Electrical stimulation of the motor cortex enhances treatment outcome in post-stroke aphasia. Brain. 2016 Apr;139(Pt 4):1152-63. doi: 10.1093/brain/aww002. Epub 2016 Feb 16. PMID 26912641
- [Background] Hesse S, Werner C, Schonhardt EM, Bardeleben A, Jenrich W, Kirker SG. Combined transcranial direct current stimulation and robot-assisted arm training in subacute stroke patients: a pilot study. Restor Neurol Neurosci. 2007;25(1):9-15. PMID 17473391
- [Background] Kang EK, Kim YK, Sohn HM, Cohen LG, Paik NJ. Improved picture naming in aphasia patients treated with cathodal tDCS to inhibit the right Broca's homologue area. Restor Neurol Neurosci. 2011;29(3):141-52. doi: 10.3233/RNN-2011-0587. PMID 21586821
- [Background] Jung IY, Lim JY, Kang EK, Sohn HM, Paik NJ. The Factors Associated with Good Responses to Speech Therapy Combined with Transcranial Direct Current Stimulation in Post-stroke Aphasic Patients. Ann Rehabil Med. 2011 Aug;35(4):460-9. doi: 10.5535/arm.2011.35.4.460. Epub 2011 Aug 31. PMID 22506160
- [Background] You DS, Kim DY, Chun MH, Jung SE, Park SJ. Cathodal transcranial direct current stimulation of the right Wernicke's area improves comprehension in subacute stroke patients. Brain Lang. 2011 Oct;119(1):1-5. doi: 10.1016/j.bandl.2011.05.002. PMID 21641021
- [Background] Turkeltaub PE, Coslett HB, Thomas AL, Faseyitan O, Benson J, Norise C, Hamilton RH. The right hemisphere is not unitary in its role in aphasia recovery. Cortex. 2012 Oct;48(9):1179-86. doi: 10.1016/j.cortex.2011.06.010. Epub 2011 Jun 30. PMID 21794852
- [Background] Naeser MA, Martin PI, Theoret H, Kobayashi M, Fregni F, Nicholas M, Tormos JM, Steven MS, Baker EH, Pascual-Leone A. TMS suppression of right pars triangularis, but not pars opercularis, improves naming in aphasia. Brain Lang. 2011 Dec;119(3):206-13. doi: 10.1016/j.bandl.2011.07.005. Epub 2011 Aug 23. PMID 21864891
- [Background] Naeser MA, Martin PI, Nicholas M, Baker EH, Seekins H, Helm-Estabrooks N, Cayer-Meade C, Kobayashi M, Theoret H, Fregni F, Tormos JM, Kurland J, Doron KW, Pascual-Leone A. Improved naming after TMS treatments in a chronic, global aphasia patient--case report. Neurocase. 2005 Jun;11(3):182-93. doi: 10.1080/13554790590944663. PMID 16006338
- [Background] Boyle M, Coelho CA. Application of semantic feature analysis as a treatment for aphasic dysnomia. Am. J. Speech Lang. Pathol. 1995;4(4):94-98
- [Background] Leonard C, Rochon E, Laird L. Treating naming impairments in aphasia: Findings from a phonological components analysis treatment. Aphasiology 2008;22(9):923-947.
- [Background] Poreisz C, Boros K, Antal A, Paulus W. Safety aspects of transcranial direct current stimulation concerning healthy subjects and patients. Brain Res Bull. 2007 May 30;72(4-6):208-14. doi: 10.1016/j.brainresbull.2007.01.004. Epub 2007 Jan 24. PMID 17452283
- [Background] Nitsche MA, Liebetanz D, Lang N, Antal A, Tergau F, Paulus W. Safety criteria for transcranial direct current stimulation (tDCS) in humans. Clin Neurophysiol. 2003 Nov;114(11):2220-2; author reply 2222-3. doi: 10.1016/s1388-2457(03)00235-9. No abstract available. PMID 14580622
- [Background] Efstratiadou EA, Papathanasiou I, Holland R, Archonti A, Hilari K. A Systematic Review of Semantic Feature Analysis Therapy Studies for Aphasia. J Speech Lang Hear Res. 2018 May 17;61(5):1261-1278. doi: 10.1044/2018_JSLHR-L-16-0330. PMID 29710193
- [Background] van Hees S, Angwin A, McMahon K, Copland D. A comparison of semantic feature analysis and phonological components analysis for the treatment of naming impairments in aphasia. Neuropsychol Rehabil. 2013;23(1):102-32. doi: 10.1080/09602011.2012.726201. Epub 2012 Oct 26. PMID 23098246

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place from August 5, 2019 through April 30, 2024 at a medical clinic and from an aphasia databank. The first participant was enrolled on December 13, 2019, and the last participant was enrolled August 11, 2023.
Pre-assignment Details: After enrollment, participants underwent screening tests to ensure behavioral criteria was met. Of the 25 enrollments, 19 met behavioral criteria and were randomized into an arm. Those who did not meet behavioral criteria did not continue in the study.
Groups:
- Phonologic-Focused Speech Therapy - Targeted tDCS First (A), Then Active Control tDCS (B): Participants will receive phonologic-focused speech therapy with targeted anodal-tDCS for 10 therapy sessions before crossing over to receive Active Control tDCS for 10 sessions.
  Transcranial Direct Current Stimulation: High-Definition-tDCS will be delivered via a battery-driven constant direct current stimulator (Soterix) using a 4x1 montage (1 central anodal electrode and 4 cathodal electrodes) arranged in a HD-cap. The current is turned on and increased in a ramplike fashion over approximately 30 seconds until reaching a strength of no more than 2mA, with a current density equal to 0.08mA/cm2. Stimulation will be maintained no longer than 20 minutes. Stimulation is either applied to the targeted or active control region, depending on the therapy cycle.
  Phonologic-Focused Speech Therapy: Participants are asked to generate or choose from a list phonologic information about a target picture.
- Phonologic-Focused Speech Therapy - Active Control tDCS First (A), Then Targeted tDCS (B): Participants will receive phonologic-focused speech therapy with active control tDCS for 10 therapy sessions before crossing over to receive target control tDCS for 10 therapy sessions.
  Transcranial Direct Current Stimulation: High-Definition-tDCS will be delivered via a battery-driven constant direct current stimulator (Soterix) using a 4x1 montage (1 central anodal electrode and 4 cathodal electrodes) arranged in a HD-cap. The current is turned on and increased in a ramplike fashion over approximately 30 seconds until reaching a strength of no more than 2mA, with a current density equal to 0.08mA/cm2. Stimulation will be maintained no longer than 20 minutes. Stimulation is either applied to the targeted or active control region, depending on the therapy cycle.
  Phonologic-Focused Speech Therapy: Participants are asked to generate or choose from a list phonologic information about a target picture.
- Semantic-Focused Speech Therapy - Targeted tDCS First (A), Then Active Control tDCS (B): Participants will receive semantic-focused speech therapy with targeted anodal-tDCS for 10 therapy sessions before crossing over to receive active-control tDCS for 10 therapy sessions.
  Transcranial Direct Current Stimulation: High-Definition-tDCS will be delivered via a battery-driven constant direct current stimulator (Soterix) using a 4x1 montage (1 central anodal electrode and 4 cathodal electrodes) arranged in a HD-cap. The current is turned on and increased in a ramplike fashion over approximately 30 seconds until reaching a strength of no more than 2mA, with a current density equal to 0.08mA/cm2. Stimulation will be maintained no longer than 20 minutes. Stimulation is either applied to the targeted or active control region, depending on the therapy cycle.
  Semantic-Focused Speech Therapy: Participants who have difficulty retrieving an object name are given hierarchical clues or asked questions about the objects function as a way of activating the semantic network for that object, leading to eventual retrieval of the target word.
- Semantic-Focused Speech Therapy Active Control tDCS First (A), Then Targeted tDCS (B): Participants will receive semantic-focused speech therapy with active control tDCS for 10 therapy sessions before crossing over to receive targted tDCS for 10 therapy sessions.
  Transcranial Direct Current Stimulation: High-Definition-tDCS will be delivered via a battery-driven constant direct current stimulator (Soterix) using a 4x1 montage (1 central anodal electrode and 4 cathodal electrodes) arranged in a HD-cap. The current is turned on and increased in a ramplike fashion over approximately 30 seconds until reaching a strength of no more than 2mA, with a current density equal to 0.08mA/cm2. Stimulation will be maintained no longer than 20 minutes. Stimulation is either applied to the targeted or active control region, depending on the therapy cycle.
  Semantic-Focused Speech Therapy: Participants who have difficulty retrieving an object name are given hierarchical clues or asked questions about the objects function as a way of activating the semantic network for that object, leading to eventual retrieval of the target word.
Period: Behavioral Assessment 1
Arm/Group | Phonologic-Focused Speech Therapy - Targeted tDCS First (A), Then Active Control tDCS (B) | Phonologic-Focused Speech Therapy - Active Control tDCS First (A), Then Targeted tDCS (B) | Semantic-Focused Speech Therapy - Targeted tDCS First (A), Then Active Control tDCS (B) | Semantic-Focused Speech Therapy Active Control tDCS First (A), Then Targeted tDCS (B)
Started | 5 | 5 | 4 | 5
Completed | 5 | 4 | 4 | 4
Not Completed | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Investigator Withdrawn | 0 | 0 | 0 | 1
Period: FMRI Session 1
Arm/Group | Phonologic-Focused Speech Therapy - Targeted tDCS First (A), Then Active Control tDCS (B) | Phonologic-Focused Speech Therapy - Active Control tDCS First (A), Then Targeted tDCS (B) | Semantic-Focused Speech Therapy - Targeted tDCS First (A), Then Active Control tDCS (B) | Semantic-Focused Speech Therapy Active Control tDCS First (A), Then Targeted tDCS (B)
Started | 5 | 4 | 4 | 4
Completed | 5 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Therapy Cycle A
Arm/Group | Phonologic-Focused Speech Therapy - Targeted tDCS First (A), Then Active Control tDCS (B) | Phonologic-Focused Speech Therapy - Active Control tDCS First (A), Then Targeted tDCS (B) | Semantic-Focused Speech Therapy - Targeted tDCS First (A), Then Active Control tDCS (B) | Semantic-Focused Speech Therapy Active Control tDCS First (A), Then Targeted tDCS (B)
Started | 5 | 4 | 4 | 4
Completed | 5 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Behavioral Assessment 2
Arm/Group | Phonologic-Focused Speech Therapy - Targeted tDCS First (A), Then Active Control tDCS (B) | Phonologic-Focused Speech Therapy - Active Control tDCS First (A), Then Targeted tDCS (B) | Semantic-Focused Speech Therapy - Targeted tDCS First (A), Then Active Control tDCS (B) | Semantic-Focused Speech Therapy Active Control tDCS First (A), Then Targeted tDCS (B)
Started | 5 | 4 | 4 | 4
Completed | 5 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: FMRI Session 2
Arm/Group | Phonologic-Focused Speech Therapy - Targeted tDCS First (A), Then Active Control tDCS (B) | Phonologic-Focused Speech Therapy - Active Control tDCS First (A), Then Targeted tDCS (B) | Semantic-Focused Speech Therapy - Targeted tDCS First (A), Then Active Control tDCS (B) | Semantic-Focused Speech Therapy Active Control tDCS First (A), Then Targeted tDCS (B)
Started | 5 | 4 | 4 | 4
Completed | 5 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Therapy Cycle B
Arm/Group | Phonologic-Focused Speech Therapy - Targeted tDCS First (A), Then Active Control tDCS (B) | Phonologic-Focused Speech Therapy - Active Control tDCS First (A), Then Targeted tDCS (B) | Semantic-Focused Speech Therapy - Targeted tDCS First (A), Then Active Control tDCS (B) | Semantic-Focused Speech Therapy Active Control tDCS First (A), Then Targeted tDCS (B)
Started | 4 (1 participant withdrew after completion of fMRI session 2, but before Therapy B stated) | 4 | 3 (1 participant withdrew after completion of fMRI session 2, but before Therapy B stated) | 4
Completed | 4 | 3 | 3 | 4
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: Behavioral Assessment 3
Arm/Group | Phonologic-Focused Speech Therapy - Targeted tDCS First (A), Then Active Control tDCS (B) | Phonologic-Focused Speech Therapy - Active Control tDCS First (A), Then Targeted tDCS (B) | Semantic-Focused Speech Therapy - Targeted tDCS First (A), Then Active Control tDCS (B) | Semantic-Focused Speech Therapy Active Control tDCS First (A), Then Targeted tDCS (B)
Started | 4 | 3 | 3 | 4
Completed | 4 | 3 | 3 | 4
Not Completed | 0 | 0 | 0 | 0
Period: FMRI Session 3
Arm/Group | Phonologic-Focused Speech Therapy - Targeted tDCS First (A), Then Active Control tDCS (B) | Phonologic-Focused Speech Therapy - Active Control tDCS First (A), Then Targeted tDCS (B) | Semantic-Focused Speech Therapy - Targeted tDCS First (A), Then Active Control tDCS (B) | Semantic-Focused Speech Therapy Active Control tDCS First (A), Then Targeted tDCS (B)
Started | 4 | 3 | 3 | 4
Completed | 4 | 3 | 3 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Behavioral Assessment 4
Arm/Group | Phonologic-Focused Speech Therapy - Targeted tDCS First (A), Then Active Control tDCS (B) | Phonologic-Focused Speech Therapy - Active Control tDCS First (A), Then Targeted tDCS (B) | Semantic-Focused Speech Therapy - Targeted tDCS First (A), Then Active Control tDCS (B) | Semantic-Focused Speech Therapy Active Control tDCS First (A), Then Targeted tDCS (B)
Started | 3 (This milestone was added after 1 participant had already completed the protocol) | 3 | 3 | 3 (This milestone was added after 1 participant had already completed the protocol)
Completed | 0 | 1 | 1 | 2
Not Completed | 3 | 2 | 2 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phonologic-Focused Speech Therapy - Targeted tDCS First, Then Active Control tDCS: Phonologic-Focused Speech Therapy - Targeted tDCS first, then Active Control tDCS.
  Participants receive phonologic speech therapy for both cycles of speech therapy. They receive targeted tDCS first, then active control tDCS second.
  Phonologic-Focused Speech Therapy: Participants are asked to generate or choose from a list phonologic information about a target picture.
- Phonologic-Focused Speech Therapy - Active Control tDCS First, Then Targeted tDCS: Phonologic-Focused Speech Therapy - Active Control tDCS first, then Targeted tDCS
  Participants receive phonologic speech therapy for both cycles of speech therapy. They receive active control tDCS first, then targeted tDCS second.
  Phonologic-Focused Speech Therapy: Participants are asked to generate or choose from a list phonologic information about a target picture.
- Semantic-Focused Speech Therapy - Targeted tDCS First, Then Active Control tDCS: Semantic-Focused Speech Therapy - Targeted tDCS first, then Active Control tDCS
  Participants receive semantic speech therapy for both cycles of speech therapy. They receive targeted tDCS first, then active control tDCS second.
  Semantic-Focused Speech Therapy: Participants who have difficulty retrieving an object name are given hierarchical clues or asked questions about the objects function as a way of activating the semantic network for that object, leading to eventual retrieval of the target word.
- Semantic-Focused Speech Therapy Active Control tDCS First, Then Targeted tDCS: Semantic-Focused Speech Therapy - Targeted tDCS first, then Active Control tDCS
  Participants receive semantic speech therapy for both cycles of speech therapy. They receive active control tDCS first, then targeted tDCS second.
  Semantic-Focused Speech Therapy: Participants who have difficulty retrieving an object name are given hierarchical clues or asked questions about the objects function as a way of activating the semantic network for that object, leading to eventual retrieval of the target word.
- Total: Total of all reporting groups
Arm/Group | Phonologic-Focused Speech Therapy - Targeted tDCS First, Then Active Control tDCS | Phonologic-Focused Speech Therapy - Active Control tDCS First, Then Targeted tDCS | Semantic-Focused Speech Therapy - Targeted tDCS First, Then Active Control tDCS | Semantic-Focused Speech Therapy Active Control tDCS First, Then Targeted tDCS | Total
Number analyzed (Participants) | 5 | 5 | 4 | 5 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 4 | 4 | 16
  >=65 years | 1 | 1 | 0 | 1 | 3
Age, Continuous [Mean (Full Range); unit: years] | 47.8 [29 to 66] | 50.8 [37 to 66] | 47.75 [40 to 57] | 59.8 [46 to 75] | 51.54 [29 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 2 | 9
  Male | 2 | 3 | 2 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 5 | 4 | 4 | 5 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 2 | 1 | 5
  White | 3 | 3 | 2 | 4 | 12
  More than one race | 2 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 4 | 5 | 19
Days Past Stroke Onset [Mean (Full Range); unit: days] — Time from stroke onset to consenting.
  days | 1525 [235 to 4487] | 1697 [121 to 3901] | 1260 [89 to 3543] | 1262 [91 to 2742] | 1436 [89 to 4487]
Years of Education [Mean (Full Range); unit: years] | 15.2 [14 to 16] | 17 [16 to 18] | 14.5 [14 to 16] | 13.2 [12 to 16] | 14.9 [12 to 18]

OUTCOME MEASURES:

1. Primary Outcome: Percent Correct on Picture Naming and Reading Tasks (Baseline on Items Was 0)
Description: Improvement on trained, untrained and untested items used during therapy. Items will consist of words and pictures that participants will name. Percent correct on lists after each therapy cycle will be the primary behavioral outcome measure (items chosen were at baseline is 0% correct).
  There were 20 pictures and 20 words in each of the trained, untrained, and untested lists. Pictures were colored photographs.
  Cycle A is the speech therapy intervention given first, Cycle B is the speech therapy intervention given second
  Cycle A Trained and Untrained lists were assessed on the last day of therapy for Cycle A Cycle A Post Trained, Untrained and Untested lists were given during Behavioral Assessment 2, approximately 10-weeks post ending Cycle A.
  Cycle B Trained and Untrained lists were assessed on the last day of therapy for Cycle B Cycle B Post Trained, Untrained and Untested lists were given during Behavioral Assessment 3, approximately 10-weeks post ending Cycle A.
Time Frame: Upon the completion of therapy cycle (a cycle consists of 10 intervention days) and 10 weeks post
Population: Cycle B participant analyzed is less than overall number to reflect participants who dropped out of the study part-way through
Measure: Mean (Standard Deviation); unit: percentage of items correct
Groups:
- Phonologic-Focused Speech Therapy - Targeted tDCS First, Then Active Control tDCS: Phonologic-Focused Speech Therapy - Targeted tDCS first, then Active Control tDCS
  Phonologic-Focused Speech Therapy: Participants are asked to generate or choose from a list phonologic information about a target picture. There are 10 therapy sessions in each cycle.
- Phonologic-Focused Speech Therapy - Active Control tDCS First, Then Targeted tDCS: Phonologic-Focused Speech Therapy - Active Control tDCS first, then Targeted tDCS
  Phonologic-Focused Speech Therapy: Participants are asked to generate or choose from a list phonologic information about a target picture. There are 10 therapy sessions in each cycle.
- Semantic-Focused Speech Therapy - Targeted tDCS First, Then Active Control tDCS: Semantic-Focused Speech Therapy - Targeted tDCS first, then Active Control tDCS
  Semantic-Focused Speech Therapy: Participants who have difficulty retrieving an object name are given hierarchical clues or asked questions about the objects function as a way of activating the semantic network for that object, leading to eventual retrieval of the target word. There are 10 therapy sessions in each cycle.
- Semantic-Focused Speech Therapy Active Control tDCS First, Then Targeted tDCS: Semantic-Focused Speech Therapy Active Control tDCS first, then Targeted tDCS
  Semantic-Focused Speech Therapy: Participants who have difficulty retrieving an object name are given hierarchical clues or asked questions about the objects function as a way of activating the semantic network for that object, leading to eventual retrieval of the target word. There are 10 speech therapy sessions in each cycle.
Arm/Group | Phonologic-Focused Speech Therapy - Targeted tDCS First, Then Active Control tDCS | Phonologic-Focused Speech Therapy - Active Control tDCS First, Then Targeted tDCS | Semantic-Focused Speech Therapy - Targeted tDCS First, Then Active Control tDCS | Semantic-Focused Speech Therapy Active Control tDCS First, Then Targeted tDCS
Number analyzed (Participants) | 5 | 5 | 4 | 5
percentage of items correct
  CycleATrainPics | 49 (47) | 72 (3) | 56 (43) | 56 (30)
  CycleATrainWord | 47 (43) | 65 (5) | 50 (13) | 42 (39)
  CycleAUntrainPic | 17 (24) | 30 (15) | 25 (24) | 10 (11)
  CycleAUntrainWord | 18 (21) | 35 (13) | 27 (15) | 27 (29)
  PostCycleATrainPic | 39 (34) | 48 (19) | 44 (32) | 30 (18)
  PostCycleATrainWord | 36 (29) | 45 (5) | 33 (13) | 45 (35)
  PostCycleAUntestPics | 18 (15) | 33 (25) | 38 (29) | 13 (18)
  PostCycleAUntestWord | 22 (19) | 27 (20) | 36 (25) | 55 (21)
  PostCycleAUntrainPic | 21 (18) | 23 (20) | 35 (13) | 18 (6)
  PostCycleAUntrainWord | 21 (15) | 33 (18) | 30 (14) | 32 (29)
  CycleBTrainPic: number analyzed (Participants) | 4 | 3 | 3 | 4
  CycleBTrainPic | 65 (46) | 64 (22) | 42 (35) | 57 (36)
  CycleBTrainWord: number analyzed (Participants) | 4 | 3 | 3 | 4
  CycleBTrainWord | 66 (31) | 65 (26) | 47 (33) | 57 (29)
  CycleBUntrainPic: number analyzed (Participants) | 4 | 3 | 3 | 4
  CycleBUntrainPic | 24 (21) | 19 (21) | 28 (32) | 19 (16)
  CycleBUntrainWord: number analyzed (Participants) | 4 | 3 | 3 | 4
  CycleBUntrainWord | 24 (19) | 24 (19) | 32 (10) | 38 (45)
  PostCycleBTrainPic: number analyzed (Participants) | 4 | 3 | 3 | 4
  PostCycleBTrainPic | 43 (37) | 21 (17) | 30 (26) | 33 (20)
  PostCycleBTrainWord: number analyzed (Participants) | 4 | 3 | 3 | 4
  PostCycleBTrainWord | 51 (34) | 40 (24) | 27 (14) | 37 (28)
  PostCycleBUntestPic: number analyzed (Participants) | 4 | 3 | 3 | 4
  PostCycleBUntestPic | 21 (20) | 19 (6) | 20 (26) | 30 (13)
  PostCycleBUntestWord: number analyzed (Participants) | 4 | 3 | 3 | 4
  PostCycleBUntestWord | 19 (19) | 16 (11) | 28 (20) | 32 (43)
  PostCycleBUntrainPic: number analyzed (Participants) | 4 | 3 | 3 | 4
  PostCycleBUntrainPic | 27 (17) | 24 (15) | 28 (24) | 29 (20)
  PostCycleBUntrainWord: number analyzed (Participants) | 4 | 3 | 3 | 4
  PostCycleBUntrainWord | 23 (18) | 28 (18) | 35 (13) | 38 (42)

2. Secondary Outcome: fMRI- Baseline
Description: Number of participants completing Rs-fMRI before therapy.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Phonologic-Focused Speech Therapy - Targeted tDCS First, Then Active Control tDCS | Phonologic-Focused Speech Therapy - Active Control tDCS First, Then Targeted tDCS | Semantic-Focused Speech Therapy - Targeted tDCS First, Then Active Control tDCS | Semantic-Focused Speech Therapy Active Control tDCS First, Then Targeted tDCS
Number analyzed (Participants) | 5 | 5 | 4 | 5
Participants | 5 | 5 | 4 | 5

3. Secondary Outcome: fMRI After Cycle A
Description: Number of participants completing Rs-fMRI after Cycle A therapy.
Time Frame: 10-weeks post Cycle A
Measure: Count of Participants; unit: Participants
Arm/Group | Phonologic-Focused Speech Therapy - Targeted tDCS First, Then Active Control tDCS | Phonologic-Focused Speech Therapy - Active Control tDCS First, Then Targeted tDCS | Semantic-Focused Speech Therapy - Targeted tDCS First, Then Active Control tDCS | Semantic-Focused Speech Therapy Active Control tDCS First, Then Targeted tDCS
Number analyzed (Participants) | 5 | 4 | 4 | 4
Participants | 5 | 4 | 4 | 4

4. Secondary Outcome: fMRI Post Cycle B
Description: Number of participants completing fMRI post Cycle B
Time Frame: 10 weeks post cycle B
Measure: Count of Participants; unit: Participants
Arm/Group | Phonologic-Focused Speech Therapy - Targeted tDCS First, Then Active Control tDCS | Phonologic-Focused Speech Therapy - Active Control tDCS First, Then Targeted tDCS | Semantic-Focused Speech Therapy - Targeted tDCS First, Then Active Control tDCS | Semantic-Focused Speech Therapy Active Control tDCS First, Then Targeted tDCS
Number analyzed (Participants) | 4 | 3 | 3 | 4
Participants | 4 | 3 | 3 | 4

5. Other Pre Specified Outcome: Performance on Outcome Measures Assessed Through the Language Battery
Description: A language battery screen assessing different language processes and providing an overall severity score (Quick Aphasia Battery or QAB) will be repeated three times (Time 1, Time 2, Time 3). Also outcomes on self-reported measures assessing confidence with speaking: Communicative Effectiveness Index (CETI), Communication Confidence Rating Scale for Aphasia (CCRSA) and overall symptoms of depression; Center for Epidemiologic Studies Short Depression Scale (CES-D-10).
  QAB = Total score range 0-10, higher scores mean less severe aphasia severity CETI= Total score range 1-100, higher scores mean better perceived communication confidence by an outside rater CCRSA = Total score range 0-100, higher scores mean more confidence in speaking ability CES-D-10= Total score range 0-30, scores >10 indicate symptoms of depression
Time Frame: 3 time points: pre-assessment, 10 weeks post-therapy cycle A and 10 weeks post-therapy cycle B
Population: Number below analyzed is different from overall number analyzed due to participants dropping out of study or self-report forms incomplete.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Phonologic-Focused Speech Therapy - Targeted tDCS First, Then Active Control tDCS: Phonologic-Focused Speech Therapy - Targeted tDCS first, then Active Control tDCS
  Phonologic-Focused Speech Therapy: Participants are asked to generate or choose from a list phonologic information about a target picture.
- Phonologic-Focused Speech Therapy - Active Control tDCS First, Then Targeted tDCS: Phonologic-Focused Speech Therapy - Active Control tDCS first, then Targeted tDCS
  Phonologic-Focused Speech Therapy: Participants are asked to generate or choose from a list phonologic information about a target picture.
- Semantic-Focused Speech Therapy - Targeted tDCS First, Then Active Control tDCS: Semantic-Focused Speech Therapy - Targeted tDCS first, then Active Control tDCS
  Semantic-Focused Speech Therapy: Participants who have difficulty retrieving an object name are given hierarchical clues or asked questions about the objects function as a way of activating the semantic network for that object, leading to eventual retrieval of the target word.
- Semantic-Focused Speech Therapy Active Control tDCS First, Then Targeted tDCS: Semantic-Focused Speech Therapy Active Control tDCS first, then Targeted tDCS
  Semantic-Focused Speech Therapy: Participants who have difficulty retrieving an object name are given hierarchical clues or asked questions about the objects function as a way of activating the semantic network for that object, leading to eventual retrieval of the target word.
Arm/Group | Phonologic-Focused Speech Therapy - Targeted tDCS First, Then Active Control tDCS | Phonologic-Focused Speech Therapy - Active Control tDCS First, Then Targeted tDCS | Semantic-Focused Speech Therapy - Targeted tDCS First, Then Active Control tDCS | Semantic-Focused Speech Therapy Active Control tDCS First, Then Targeted tDCS
Number analyzed (Participants) | 5 | 4 | 4 | 4
score on a scale
  QAB total T1 | 6 (3) | 6 (1) | 7 (2) | 7 (2)
  QAB total T2: number analyzed (Participants) | 5 | 3 | 4 | 4
  QAB total T2 | 5 (4) | 7 (1) | 7 (2) | 7 (2)
  QAB total T3: number analyzed (Participants) | 4 | 3 | 3 | 4
  QAB total T3 | 6 (3) | 7 (1) | 6 (0) | 7 (3)
  CETI T1: number analyzed (Participants) | 4 | 3 | 4 | 4
  CETI T1 | 66 (38) | 100 (32) | 78 (28) | 102 (37)
  CETI T2: number analyzed (Participants) | 3 | 2 | 4 | 4
  CETI T2 | 82 (61) | 122 (13) | 81 (27) | 104 (30)
  CETI T3: number analyzed (Participants) | 3 | 2 | 3 | 4
  CETI T3 | 85 (60) | 117 (15) | 83 (17) | 108 (21)
  CCRSA T1: number analyzed (Participants) | 4 | 3 | 4 | 4
  CCRSA T1 | 50 (20) | 68 (29) | 56 (23) | 66 (26)
  CCRSA T2: number analyzed (Participants) | 4 | 3 | 4 | 4
  CCRSA T2 | 51 (24) | 77 (17) | 66 (22) | 63 (15)
  CCRSA T3: number analyzed (Participants) | 4 | 3 | 3 | 4
  CCRSA T3 | 61 (20) | 78 (9) | 71 (10) | 71 (11)
  CESD T1: number analyzed (Participants) | 4 | 3 | 4 | 4
  CESD T1 | 13 (8) | 7 (8) | 13 (13) | 4 (5)
  CESD T2: number analyzed (Participants) | 4 | 3 | 4 | 4
  CESD T2 | 8 (4) | 5 (6) | 8 (6) | 8 (7)
  CESD T3: number analyzed (Participants) | 4 | 3 | 3 | 4
  CESD T3 | 8 (4) | 8 (7) | 6 (4) | 5 (9)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the first day of intervention until up to six months after the last day of intervention.
Description: Adverse event data were collected systematically on the last day of each treatment period.
  Non-systematic adverse event data were also collected during a participant's study duration starting from the first study activity until up to 6 months post treatment 2.
Groups:
- Phonologic-Focused Speech Therapy - Targeted tDCS: Phonologic-Focused Speech Therapy - Targeted tDCS
  Phonologic-Focused Speech Therapy: Participants are asked to generate or choose from a list phonologic information about a target picture.
- Phonologic-Focused Speech Therapy - Active Control tDCS: Phonologic-Focused Speech Therapy - Active Control tDCS
  Phonologic-Focused Speech Therapy: Participants are asked to generate or choose from a list phonologic information about a target picture.
- Semantic-Focused Speech Therapy - Targeted tDCS: Semantic-Focused Speech Therapy - Targeted tDCS
  Semantic-Focused Speech Therapy: Participants who have difficulty retrieving an object name are given hierarchical clues or asked questions about the objects function as a way of activating the semantic network for that object, leading to eventual retrieval of the target word.
- Semantic-Focused Speech Therapy - Active Control tDCS: Semantic-Focused Speech Therapy Active Control tDCS
  Semantic-Focused Speech Therapy: Participants who have difficulty retrieving an object name are given hierarchical clues or asked questions about the objects function as a way of activating the semantic network for that object, leading to eventual retrieval of the target word.
Arm/Group | Phonologic-Focused Speech Therapy - Targeted tDCS | Phonologic-Focused Speech Therapy - Active Control tDCS | Semantic-Focused Speech Therapy - Targeted tDCS | Semantic-Focused Speech Therapy - Active Control tDCS
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 1/8 | 0/8 | 3/8 | 2/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phonologic-Focused Speech Therapy - Targeted tDCS (N=8) | Phonologic-Focused Speech Therapy - Active Control tDCS (N=8) | Semantic-Focused Speech Therapy - Targeted tDCS (N=8) | Semantic-Focused Speech Therapy - Active Control tDCS (N=7)
Headache (General disorders) | 0 | 0 | 1 | 0
Skin Discomfort (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 2 — Discomfort at stimulation site

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-05): https://cdn.clinicaltrials.gov/large-docs/13/NCT04166513/Prot_SAP_002.pdf
  • Informed Consent Form (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/13/NCT04166513/ICF_001.pdf